CLINICAL TRIAL: NCT03382158
Title: International Pleuropulmonary Blastoma/DICER1 Registry (for PPB, DICER1 and Associated Conditions)
Brief Title: International PPB/DICER1 Registry
Status: Recruiting | Type: Observational
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Collaborators: Washington University School of Medicine (Other); ResourcePath, LLC (Unknown); University of Cambridge (Other); Emory University (Other); Dana-Farber Cancer Institute (Other); Phoenix Children's Hospital (Other); Allina Health System (Other); University of California, San Francisco (Other); M.D. Anderson Cancer Center (Other); UC Davis Children's Hospital (Unknown); KK Women's and Children's Hospital (Other Government); Louisiana State University Health Sciences Center Shreveport (Other); Children's Healthcare of Atlanta (Other); Dayton Children's Hospital (Other); Akron Children's Hospital (Other); Starship Children's Hospital of New Zealand (Unknown); Beijing Children's Hospital (Other); Bronson Methodist Hospital (Unknown); Rutgers Cancer Institute of New Jersey (Other); Children's Hospital of Los Angeles (CHLA) (Unknown); Children's Hospital of Philadelphia (Other); Cincinnati Children's Hospital Medical Center (CCHMC) (Unknown); Connecticut Children's Medical Center (Other); Federal Scientific Clinical Centre of Pediatric Hematology, Oncology and Immunology named after Dmitry Rogache (Other); Driscoll Children's Hospital (Other); Hannover Medical School (Other); Jewish General Hospital (Other); Kaiser Permanente (Other); King Faisal Specialist Hospital & Research Center (Other); Kingston Health Sciences Centre (Other); Massachusetts General Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); National Institutes of Health (NIH) (NIH); Royal Perth Hospital (Other); Princess Margaret Hospital for Children (Other); Prisma Health-Upstate (Other); Roswell Park Cancer Institute (Other); The Hospital for Sick Children (SickKids) (Unknown); St. Jude Children's Research Hospital (Other); Huntsman Cancer Institute/ University of Utah (Unknown); University of Virginia (Other); University of Texas Southwestern Medical Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: FDAAA
Record Dates: First submitted 2017-10-11; First posted 2017-12-22 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Pleuropulmonary Blastoma; Sertoli-Leydig Cell Tumor; DICER1 Syndrome; Cystic Nephroma; Wilms Tumor; Pineoblastoma; Renal Sarcoma; Nodular Hyperplasia of Thyroid; Nasal Chondromesenchymal Hamartoma; Ciliary Body Medulloepithelioma; Neuroblastoma; Pituitary Cancer; Embryonal Rhabdomyosarcoma; Ovarian Sarcoma; Gynandroblastoma; Thyroid Carcinoma; Embryonal Rhabdomyosarcoma of Vagina (Diagnosis); Embryonal Rhabdomyosarcoma of Uterus (Diagnosis); Embryonal Rhabdomyosarcoma of Cervix
Keywords: pleuropulmonary blastoma; PPB; DICER1; SLCT; Sertoli-Leydig Cell Tumor; Cystic Nephroma; CN; DICER1 mutation; DICER1 syndrome; Wilms Tumor; Pineoblastoma; Renal Sarcoma; ASK; Nodular Hyperplasia of Thyroid; Thyroid Nodules; Thyroid Carcinoma; Nasal Chondromesenchymal Hamartoma; NCMH; Ciliary Body Medulloepithelioma; CBME; Neuroblastoma; Pituitary Cancer; Embryonal Rhabdomyosarcoma; ERMS; Ovarian Sarcoma; Gynandroblastoma; Peritoneal PPB; pPPB; multinodular goiter; PPB Type I; PPB Type II; PPB Type III; PPB Type Ir
MeSH Terms: conditions — Pleuropulmonary blastoma; Sertoli-Leydig Cell Tumor; Wilms Tumor; Pinealoma; Goiter, Nodular; Neuroblastoma; Pituitary Neoplasms; Rhabdomyosarcoma, Embryonal; Sex Cord-Gonadal Stromal Tumors; Thyroid Neoplasms; Disease; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tumor tissue, blood, urine, and cerebral spinal fluid (the latter only if a lumbar puncture is performed for clinical purposes) can be collected from enrolled individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Type I PPB: Type I PPB is an early manifestation of this malignant disease, cured in some cases by surgery. Surgical guidelines are presented. It is unknown whether adjuvant chemotherapy improves cure rates for individuals with Type I PPB. If the treating physicians select adjuvant chemotherapy treatment, chemotherapy options include a 22-week regimen: 4 courses of vincristine, actinomycin D and cyclophosphamide (VAC) followed by 3 courses of vincristine and actinomycin D (VA). Therapy decisions are the responsibility of the treating institution.
- Types II and III PPB: Types II and III PPB are aggressive sarcomas. Surgery and chemotherapy are necessary in all cases. Surgical guidelines are presented. Many children with Types II or III PPB receive a single-arm multi-agent chemotherapy neo-adjuvant/adjuvant regimen of IVADo (ifosfamide, vincristine, actinomycin, doxorubicin) for 36 weeks. Second and possible 3rd look surgery may be considered for local control. Radiation therapy may be considered. Specific therapy decisions are the responsibility of the treating institution.
- Type Ir PPB: Type Ir (regressed) PPB is a unique, purely cystic tumor which lacks a primitive cell component. The International PPB/DICER1 Registry will enroll and follow participants with Type Ir PPB, regardless of age.
- DICER1 Gene or Cond Assoc with DICER1: PPB and the associated conditions found in PPB families suggest a familial tendency to formation of tumors. The International PPB/DICER1 Registry for PPB, DICER1 and Associated Conditions study will enroll and follow participants who have the DICER1 gene mutations or conditions associated with PPB or DICER1.

SUMMARY:
Pleuropulmonary blastoma (PPB) is a rare malignant neoplasm of the lung presenting in early childhood. Type I PPB is a purely cystic lesion, Type II is a partially cystic, partially solid tumor, Type III is a completely solid tumor. Treatment of children with PPB is at the discretion of the treating institution. This study builds off of the 2009 study and will also seek to enroll individuals with DICER1-associated conditions, some of whom may present only with the DICER1 gene mutation, which will help the Registry understand how these tumors and conditions develop, their clinical course and the most effective treatments.

DETAILED DESCRIPTION:
PPB is a rare cancer of the lung presenting in early childhood, mostly commonly from birth to age ~72 months. PPB occurs within the lung or between the lung and the chest wall. There are three primary forms of PPB called Types I, II, and III PPB. PPB is related to an underlying change/mutation in a gene called DICER1 which impacts gene expression and cell growth. DICER1 mutations may also lead to the development of other tumors in children and adults.

The International PPB/DICER1 Registry offers information based on previous data from Registry participants and the medical literature and collaborative efforts with international rare tumor groups.

Retrospective and real-time central pathology review is encouraged. Therapy decisions remain at the discretion of the treating institution.

Children with Type I PPB require surgery and sometimes chemotherapy. Therapy decisions are the responsibility of the treating institution. Surgical guidelines are presented. It is unknown whether adjuvant chemotherapy improves cure rates for Type I PPB patients. Chemotherapy options include a 22-week regimen: 4 courses of vincristine, actinomycin D and cyclophosphamide (VAC) followed by 3 courses of vincristine and actinomycin D (VA).

Children with Types II and III PPB, require surgery, chemotherapy and sometimes radiation therapy. Many children with Types II or III PPB receive a single-arm multi-agent chemotherapy neo-adjuvant/adjuvant regimen of IVADo (ifosfamide, vincristine, actinomycin, doxorubicin) for 36 weeks. Second and possible 3rd look surgery may be considered for local control. Radiation therapy may be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Known or suspected PPB or related thoracic tumor
2. Known or suspected sex-cord stromal tumor including Sertoli-Leydig cell tumor and gynandroblastoma (males or females)
3. Other known or suspected DICER1-related condition including ovarian sarcoma, cystic nephroma, renal sarcoma, pineoblastoma, pituitary blastoma, nasal chondromesenchymal hamartoma, ciliary body medulloepithelioma and others
4. Individuals with known or suspected DICER1 pathogenic variation regardless of whether they have an established DICER1-associated condition
5. Informed consent by patient/ or parent/guardian (also, where appropriate: assent and HIPAA consent)

Exclusion criteria:

Absence of appropriate consent for Registry participation

Ages: 0 Minutes to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. For those with PPB: PPB primarily affects children so their participation is required.
  2. For those with DICER1-associated conditions: There's a wide array of conditions associated with DICER1, that occur at a variety of ages, from the development of cysts in utero, to lung cysts and thyroid disease noted in grandparents.
  3. The Investigators are aware that many individuals with PPB, and with conditions associated with DICER1, come from countries outside of the U.S. To exclude individuals outside the US, minority groups and non-English speaking groups would be a disservice to eligible patients and healthcare providers and would limit the sample size of this rare cancer study.
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Estimated)
Dates: Start 2016-12-06 (Actual); Primary Completion 2030-12-06 (Estimated); Study Completion 2035-12-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 7 years
  The primary endpoint for statistical analysis will be time from start treatment to an event, defined as the occurrence of progression or recurrence of PPB, occurrence of a second malignant neoplasm, or death from any cause that is at least possibly related to the original disease or treatment.

SECONDARY OUTCOMES:
Overall response to chemotherapy | 7 years
  The investigators will assess overall response to chemotherapy among participants with radiographically measurable tumor following initial surgery or biopsy.
Overall survival | 7 years
  The investigators will assess overall survival and time to death from any cause among participants.
Quality of life outcomes in individuals diagnosed with PPB. | 7 years
  Chemotherapy and surgery may have adverse effects on the quality of life outcomes. Multiple factors may impact quality of life for participants.This study will allow the investigators to assess the quality of life outcomes in participants with DICER1-related tumors and will compare outcomes to those with more common childhood cancers.
Cardiac outcomes in individuals diagnosed with PPB. | 7 years
  Chemotherapy and surgery may have adverse effects on cardiac outcomes. This study will allow the investigators to assess the cardiac outcomes as measured by ejection fraction and shortening fraction via echocardiogram of participants with DICER1-related tumors, and compare outcomes to those with more common childhood cancers.
Pulmonary function testing results in individuals diagnosed with PPB | 7 years
  Chemotherapy and surgery may have adverse effects on pulmonary outcomes. This study will allow the investigators to assess the pulmonary outcome of participants as ascertained by pulmonary function testing (forced vital capacity (FVC), FEV1(forced expiratory volume in 1 second)/FVC) with DICER1-related tumors, and compare outcomes to those with more common childhood cancers.
Incidence of neoplasms in individuals with DICER1-related conditions or germline DICER1 variants. mutation. | 7 years
  This protocol will include individuals with germline DICER1 mutations and will calculate incidence rates of specific neoplasms in this population

CONTACTS AND LOCATIONS:
Overall Officials: Kris Ann P Schultz, MD, Principal Investigator — Children's Minnesota
Locations (1):
- Children's Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill DA, Ivanovich J, Priest JR, Gurnett CA, Dehner LP, Desruisseau D, Jarzembowski JA, Wikenheiser-Brokamp KA, Suarez BK, Whelan AJ, Williams G, Bracamontes D, Messinger Y, Goodfellow PJ. DICER1 mutations in familial pleuropulmonary blastoma. Science. 2009 Aug 21;325(5943):965. doi: 10.1126/science.1174334. Epub 2009 Jun 25. PMID 19556464
- [Background] Messinger YH, Stewart DR, Priest JR, Williams GM, Harris AK, Schultz KA, Yang J, Doros L, Rosenberg PS, Hill DA, Dehner LP. Pleuropulmonary blastoma: a report on 350 central pathology-confirmed pleuropulmonary blastoma cases by the International Pleuropulmonary Blastoma Registry. Cancer. 2015 Jan 15;121(2):276-85. doi: 10.1002/cncr.29032. Epub 2014 Sep 10. PMID 25209242
- [Background] Vasta LM, McMaster ML, Harney LA, Ling A, Kim J, Harris AK, Carr AG, Damrauer SM, Rader DJ, Kember RL, Kanetsky PA, Nathanson KL, Pyle LC, Greene MH, Schultz KA, Stewart DR; Regeneron Genetics Center (RGC) Research Team. Lack of pathogenic germline DICER1 variants in males with testicular germ-cell tumors. Cancer Genet. 2020 Oct;248-249:49-56. doi: 10.1016/j.cancergen.2020.10.002. Epub 2020 Oct 24. PMID 33158809
- [Background] Schneider KW, Cost NG, Schultz KAP, Svihovec S, Suttman A. Germline predisposition to genitourinary rhabdomyosarcoma. Transl Androl Urol. 2020 Oct;9(5):2430-2440. doi: 10.21037/tau-20-76. PMID 33209717
- [Background] Bisogno G, Sarnacki S, Stachowicz-Stencel T, Minard Colin V, Ferrari A, Godzinski J, Gauthier Villars M, Bien E, Hameury F, Helfre S, Schneider DT, Reguerre Y, Lopez Almaraz R, Janic D, Cesen M, Kolenova A, Rascon J, Martinova K, Cosnarovici R, Pourtsidis A, Ben Ami T, Roganovic J, Koscielniak E, Schultz KAP, Brecht IB, Orbach D. Pleuropulmonary blastoma in children and adolescents: The EXPeRT/PARTNER diagnostic and therapeutic recommendations. Pediatr Blood Cancer. 2021 Jun;68 Suppl 4(Suppl 4):e29045. doi: 10.1002/pbc.29045. Epub 2021 Apr 7. PMID 33826235
- [Background] Kebudi R, Dural O, Bay SB, Gorgun O, Onder S, Bilgic B, Yilmaz I, Iribas A, Arndt CA, Harris AK, Field A, Schultz KAP, Hill DA. Childhood Rhabdomyosarcoma of the Female Genital Tract: Association with Pathogenic DICER1 Variation, Clinicopathological Features, and Outcomes. J Pediatr Adolesc Gynecol. 2021 Aug;34(4):449-453. doi: 10.1016/j.jpag.2021.01.011. Epub 2021 Jan 20. PMID 33484847
- [Background] Golmard L, Vasta LM, Duflos V, Corsini C, Dubois d'Enghien C, McMaster ML, Harney LA, Carr AG, Ling A, Dijoud F, Gauthier A, Miettinen M, Cost NG, Gauthier-Villars M, Orbach D, Irtan S, Haouy S, Schultz KA, Stoppa-Lyonnet D, Coupier I, Stewart DR, Sirvent N. Testicular Sertoli cell tumour and potentially testicular Leydig cell tumour are features of DICER1 syndrome. J Med Genet. 2022 Apr;59(4):346-350. doi: 10.1136/jmedgenet-2020-107434. Epub 2021 Mar 29. PMID 33782093
- [Background] Schneider DT, Orbach D, Ben-Ami T, Bien E, Bisogno G, Brecht IB, Cecchetto G, Ferrari A, Godzinski J, Janic D, Lopez Almaraz R, Pourtsidis A, Roganovic J, Schultz KAP, Stachowicz-Stencel T, Fresneau B. Consensus recommendations from the EXPeRT/PARTNER groups for the diagnosis and therapy of sex cord stromal tumors in children and adolescents. Pediatr Blood Cancer. 2021 Jun;68 Suppl 4:e29017. doi: 10.1002/pbc.29017. Epub 2021 Mar 24. PMID 33760357
- [Background] Caron CP, Turcotte B, Pelland-Marcotte MC, Schultz KAP, Harvey I, Bolduc S. Case - Bilateral and recurrent pediatric cystic nephroma associated with DICER1 mutation. Can Urol Assoc J. 2021 May;15(5):E290-E292. doi: 10.5489/cuaj.6836. No abstract available. PMID 33119505
- [Background] Vasta LM, Khan NE, Higgs CP, Harney LA, Carr AG, Harris AK, Schultz KAP, McMaster ML, Stewart DR. Hematologic indices in individuals with pathogenic germline DICER1 variants. Blood Adv. 2021 Jan 12;5(1):216-223. doi: 10.1182/bloodadvances.2020002651. PMID 33570641
- [Background] Ferguson MJ, Ivanovich J, Stansell P, Vik TA, Helvie AE, Schmitt MR, Schultz KA, Dehner LP, Renbarger JL, Marshall MS. Previously unreported somatic variants in two patients with pleuropulmonary blastoma with metastatic brain recurrence. Pediatr Blood Cancer. 2021 May;68(5):e28825. doi: 10.1002/pbc.28825. Epub 2020 Nov 30. No abstract available. PMID 33258270
- [Background] Dural O, Kebudi R, Yavuz E, Yilmaz I, Buyukkapu Bay S, Schultz KAP, Hill DA. DICER1-Related Embryonal Rhabdomyosarcoma of the Uterine Corpus in a Prepubertal Girl. J Pediatr Adolesc Gynecol. 2020 Apr;33(2):173-176. doi: 10.1016/j.jpag.2019.12.002. Epub 2019 Dec 12. PMID 31838154
- [Background] Gonzalez IA, Mallinger P, Watson D, Harris AK, Messinger YH, Schultz KAP, Field A, Hill DA, Dehner LP. Expression of p53 is significantly associated with recurrence-free survival and overall survival in pleuropulmonary blastoma (PPB): a report from the International Pleuropulmonary Blastoma/DICER1 Registry. Mod Pathol. 2021 Jun;34(6):1104-1115. doi: 10.1038/s41379-021-00735-8. Epub 2021 Feb 26. PMID 33637876
- [Background] Schultz KAP, Williams GM, Kamihara J, Stewart DR, Harris AK, Bauer AJ, Turner J, Shah R, Schneider K, Schneider KW, Carr AG, Harney LA, Baldinger S, Frazier AL, Orbach D, Schneider DT, Malkin D, Dehner LP, Messinger YH, Hill DA. DICER1 and Associated Conditions: Identification of At-risk Individuals and Recommended Surveillance Strategies. Clin Cancer Res. 2018 May 15;24(10):2251-2261. doi: 10.1158/1078-0432.CCR-17-3089. Epub 2018 Jan 17. PMID 29343557
- [Background] Schultz KAP, Rednam SP, Kamihara J, Doros L, Achatz MI, Wasserman JD, Diller LR, Brugieres L, Druker H, Schneider KA, McGee RB, Foulkes WD. PTEN, DICER1, FH, and Their Associated Tumor Susceptibility Syndromes: Clinical Features, Genetics, and Surveillance Recommendations in Childhood. Clin Cancer Res. 2017 Jun 15;23(12):e76-e82. doi: 10.1158/1078-0432.CCR-17-0629. PMID 28620008
- [Background] Schultz KAP, Stewart DR, Kamihara J, Bauer AJ, Merideth MA, Stratton P, Huryn LA, Harris AK, Doros L, Field A, Carr AG, Dehner LP, Messinger Y, Hill DA. DICER1 Tumor Predisposition. 2014 Apr 24 [updated 2020 Apr 30]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK196157/ PMID 24761742
- [Background] Li BK, Vasiljevic A, Dufour C, Yao F, Ho BLB, Lu M, Hwang EI, Gururangan S, Hansford JR, Fouladi M, Nobusawa S, Laquerriere A, Delisle MB, Fangusaro J, Forest F, Toledano H, Solano-Paez P, Leary S, Birks D, Hoffman LM, Szathmari A, Faure-Conter C, Fan X, Catchpoole D, Zhou L, Schultz KAP, Ichimura K, Gauchotte G, Jabado N, Jones C, Loussouarn D, Mokhtari K, Rousseau A, Ziegler DS, Tanaka S, Pomeroy SL, Gajjar A, Ramaswamy V, Hawkins C, Grundy RG, Hill DA, Bouffet E, Huang A, Jouvet A. Pineoblastoma segregates into molecular sub-groups with distinct clinico-pathologic features: a Rare Brain Tumor Consortium registry study. Acta Neuropathol. 2020 Feb;139(2):223-241. doi: 10.1007/s00401-019-02111-y. Epub 2019 Dec 9. PMID 31820118
- [Background] Stewart DR, Best AF, Williams GM, Harney LA, Carr AG, Harris AK, Kratz CP, Dehner LP, Messinger YH, Rosenberg PS, Hill DA, Schultz KAP. Neoplasm Risk Among Individuals With a Pathogenic Germline Variant in DICER1. J Clin Oncol. 2019 Mar 10;37(8):668-676. doi: 10.1200/JCO.2018.78.4678. Epub 2019 Feb 4. PMID 30715996
- [Background] Kamihara J, Paulson V, Breen MA, Laetsch TW, Rakheja D, Shulman DS, Schoettler ML, Clinton CM, Ward A, Reidy D, Pinches RS, Weiser DA, Mullen EA, Schienda J, Meyers PA, DuBois SG, Nowak JA, Foulkes WD, Schultz KAP, Janeway KA, Vargas SO, Church AJ. DICER1-associated central nervous system sarcoma in children: comprehensive clinicopathologic and genetic analysis of a newly described rare tumor. Mod Pathol. 2020 Oct;33(10):1910-1921. doi: 10.1038/s41379-020-0516-1. Epub 2020 Apr 14. PMID 32291395
- [Background] Kalish JM, Doros L, Helman LJ, Hennekam RC, Kuiper RP, Maas SM, Maher ER, Nichols KE, Plon SE, Porter CC, Rednam S, Schultz KAP, States LJ, Tomlinson GE, Zelley K, Druley TE. Surveillance Recommendations for Children with Overgrowth Syndromes and Predisposition to Wilms Tumors and Hepatoblastoma. Clin Cancer Res. 2017 Jul 1;23(13):e115-e122. doi: 10.1158/1078-0432.CCR-17-0710. PMID 28674120
- [Background] Kim J, Schultz KAP, Hill DA, Stewart DR. The prevalence of germline DICER1 pathogenic variation in cancer populations. Mol Genet Genomic Med. 2019 Mar;7(3):e555. doi: 10.1002/mgg3.555. Epub 2019 Jan 22. PMID 30672147
- [Background] Nakano Y, Gatell SP, Schultz KAP, Carrillo TM, Fujisaki H, Okada K, Horiike M, Nakamura T, Watanabe Y, Matsusaka Y, Sakamoto H, Fukushima H, Inoue T, Williams GM, Hill DA, Hara J. Successful treatment of metastatic cerebral recurrence of pleuropulmonary blastoma. Pediatr Blood Cancer. 2019 May;66(5):e27628. doi: 10.1002/pbc.27628. Epub 2019 Jan 24. PMID 30677214
- [Background] Bauer AJ, Stewart DR, Kamihara J, Harris AK, Turner J, Shah R, Schneider KW, Schneider K, Carr AG, Harney LA, Frazier AL, Orbach D, Schneider DT, Malkin D, Dehner LP, Messinger YH, Hill DA, Schultz KAP. DICER1 and Associated Conditions: Identification of At-risk Individuals and Recommended Surveillance Strategies-Response. Clin Cancer Res. 2019 Mar 1;25(5):1689-1690. doi: 10.1158/1078-0432.CCR-18-3495. No abstract available. PMID 30824630
- [Background] Nakano Y, Hasegawa D, Stewart DR, Schultz KAP, Harris AK, Hirato J, Uemura S, Tamura A, Saito A, Kawamura A, Yoshida M, Yamasaki K, Yamashita S, Ushijima T, Kosaka Y, Ichimura K, Dehner LP, Hill DA. Presacral malignant teratoid neoplasm in association with pathogenic DICER1 variation. Mod Pathol. 2019 Dec;32(12):1744-1750. doi: 10.1038/s41379-019-0319-4. Epub 2019 Jul 11. PMID 31296931
- [Background] Merideth MA, Harney LA, Vyas N, Bachi A, Carr AG, Hill DA, Dehner LP, Schultz KAP, Stewart DR, Stratton P. Gynecologic and reproductive health in patients with pathogenic germline variants in DICER1. Gynecol Oncol. 2020 Mar;156(3):647-653. doi: 10.1016/j.ygyno.2019.12.037. Epub 2020 Jan 15. PMID 31952842
- [Background] Schultz KAP, Nelson A, Harris AK, Finch M, Field A, Jarzembowski JA, Wilhelm M, Mize W, Kreiger P, Conard K, Walter A, Olson T, Mitchell S, Runco DV, Bechtel A, Klawinski D, Bradfield S, Gettinger K, Stewart DR, Messinger Y, Dehner LP, Ashley Hill D. Pleuropulmonary blastoma-like peritoneal sarcoma: a newly described malignancy associated with biallelic DICER1 pathogenic variation. Mod Pathol. 2020 Oct;33(10):1922-1929. doi: 10.1038/s41379-020-0558-4. Epub 2020 May 15. PMID 32415267
- [Background] Khan NE, Ling A, Raske ME, Harney LA, Carr AG, Field A, Harris AK, Williams GM, Dehner LP, Messinger YH, Hill DA, Schultz KAP, Stewart DR. Structural renal abnormalities in the DICER1 syndrome: a family-based cohort study. Pediatr Nephrol. 2018 Dec;33(12):2281-2288. doi: 10.1007/s00467-018-4040-1. Epub 2018 Sep 3. PMID 30178239
- [Background] Huryn LA, Turriff A, Harney LA, Carr AG, Chevez-Barrios P, Gombos DS, Ram R, Hufnagel RB, Hill DA, Zein WM, Schultz KAP, Bishop R, Stewart DR. DICER1 Syndrome: Characterization of the Ocular Phenotype in a Family-Based Cohort Study. Ophthalmology. 2019 Feb;126(2):296-304. doi: 10.1016/j.ophtha.2018.09.038. Epub 2018 Oct 17. PMID 30339877
- [Background] Khan NE, Bauer AJ, Doros L, Schultz KA, Decastro RM, Harney LA, Kase RG, Carr AG, Harris AK, Williams GM, Dehner LP, Messinger YH, Stewart DR. Macrocephaly associated with the DICER1 syndrome. Genet Med. 2017 Feb;19(2):244-248. doi: 10.1038/gim.2016.83. Epub 2016 Jul 21. PMID 27441995
- [Background] Dehner LP, Hill DA, Stewart DR, Schultz KAP. Reply: pleuropulmonary blastoma-like peritoneal sarcoma and DICER1-associated sarcomas: toward a unified nomenclature. Mod Pathol. 2021 Jun;34(6):1229-1230. doi: 10.1038/s41379-021-00810-0. Epub 2021 Apr 19. No abstract available. PMID 33875804
- [Background] Mirshahi UL, Kim J, Best AF, Chen ZE, Hu Y, Haley JS, Golden A, Stahl R, Manickam K, Carr AG, Harney LA, Field A, Hatton J, Schultz KAP, Bauer AJ, Hill DA, Rosenberg PS, Murray MF, Carey DJ, Stewart DR. A Genome-First Approach to Characterize DICER1 Pathogenic Variant Prevalence, Penetrance, and Phenotype. JAMA Netw Open. 2021 Feb 1;4(2):e210112. doi: 10.1001/jamanetworkopen.2021.0112. PMID 33630087
- [Background] Gonzalez IA, Stewart DR, Schultz KAP, Field AP, Hill DA, Dehner LP. DICER1 tumor predisposition syndrome: an evolving story initiated with the pleuropulmonary blastoma. Mod Pathol. 2022 Jan;35(1):4-22. doi: 10.1038/s41379-021-00905-8. Epub 2021 Oct 1. PMID 34599283
- [Background] Terry W, Carlisle EM, Mallinger P, Nelson AT, Gordon D, Messinger YH, Field A, Dehner LP, Hill DA, Schultz KAP. Thoracic Sertoli-Leydig cell tumor: An alternative type of pleuropulmonary blastoma associated with DICER1 variation. Pediatr Blood Cancer. 2021 Nov;68(11):e29284. doi: 10.1002/pbc.29284. Epub 2021 Aug 16. PMID 34398502
- See also: International Pleuropulmonary Blastoma (PPB)/DICER1 Registry web site — http://www.PPBregistry.org